CLINICAL TRIAL: NCT01621659
Title: Multidisciplinary Team IntervenTion in CArdio-ONcology
Brief Title: Multidisciplinary Team IntervenTion in CArdio-ONcology (TITAN Study)
Acronym: TITAN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TITAN 102
Record Dates: First submitted 2012-06-04; First posted 2012-06-18 (Estimated); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: multidisciplinary team; exercise; nutrition; cardiology; physiotherapy; imaging
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Methods; Nutrition Assessment; Counseling

STUDY DESIGN:
Intervention Model Description: Supportive care intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- multidisciplinary team intervention (Experimental): Intervention arm receives regular assessments and treatments from cardiology team, clinical nutrition, pharmacist, exercise physiologist and physiotherapist
  Interventions: Behavioral: Multidisciplinary team intervention
- Observational arm (No Intervention): Participants randomized to observational arm will receive usual care.

INTERVENTIONS:
Behavioral: Multidisciplinary team intervention — Intervention arm receives regular assessments and treatments from cardiology team, clinical nutrition, pharmacist, exercise physiologist and physiotherapist
  Other Names: cardiology assessment and intervention; nutritional assessment and intervention; exercise assessment and training; pharmacist assessment and counseling; physiotherapy assessment and training
  Arms: multidisciplinary team intervention

SUMMARY:
People with breast cancer often experience many short and long-term side effects as a result of both the cancer and the necessary treatments.

Receiving extra assessments and care from teams of multiple health professionals has been shown to be helpful for people with other health problems, such as heart disease. These 'multidisciplinary' teams may include nurses, doctors, pharmacists, dietitians, exercise therapists, counselors, and other specialists. Currently, the investigators do not know if receiving extra assessments from a multidisciplinary team is helpful for people receiving cancer treatment.

In this study, the investigators hope to learn the effect of extra assessments and early interventions from teams of health care professionals in people diagnosed with cancer, during and after the treatment period.

After initial assessments, participants will be randomized to multidisciplinary team intervention or usual care.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed malignancy (breast or lymphoma);
* scheduled to receive anthracycline and/or trastuzumab-based chemotherapy;
* age ≥ 18 years;
* willing to attend follow-up visits.

Exclusion Criteria:

* physical disability preventing exercise testing or DEXA scan;
* psychiatric disease or disorder precluding informed consent;
* participation in other cardiotoxicity or exercise intervention study;
* contraindication to anti-cancer therapy, including known heart failure, cardiomyopathy, or baseline LVEF < 50%;
* previous anthracycline or trastuzumab-based therapy;
* previous radiotherapy to thorax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2018-05-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
cardiac MRI | change from baseline to 12 months
  left ventricular ejection fraction (LVEF)

SECONDARY OUTCOMES:
serum biomarkers | change from baseline to 12 months
  percent change in established biomarkers (troponin, BNP)

OTHER OUTCOMES:
multidisciplinary team interventions | change from baseline to 12 months
  nutrition, exercise, physiotherapy interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Kirkham AA, Mackey JR, Thompson RB, Haykowsky MJ, Oudit GY, McNeely M, Coulden R, Stickland MK, Baracos VE, Dyck JRB, Haennel R, Pituskin E, Paterson DI. TITAN Trial: A Randomized Controlled Trial of a Cardiac Rehabilitation Care Model in Breast Cancer. JACC Adv. 2023 Jul 27;2(6):100424. doi: 10.1016/j.jacadv.2023.100424. eCollection 2023 Aug. PMID 38939428
- [Derived] Maayah ZH, Ferdaoussi M, Boukouris AE, Takahara S, Das SK, Khairy M, Mackey JR, Pituskin E, Sutendra G, Paterson DI, Dyck JRB. Endothelin Receptor Blocker Reverses Breast Cancer-Induced Cardiac Remodeling. JACC CardioOncol. 2023 May 2;5(5):686-700. doi: 10.1016/j.jaccao.2023.02.004. eCollection 2023 Oct. PMID 37969640
- [Derived] Pituskin E, Haykowsky M, McNeely M, Mackey J, Chua N, Paterson I. Rationale and design of the multidisciplinary team IntervenTion in cArdio-oNcology study (TITAN). BMC Cancer. 2016 Sep 15;16(1):733. doi: 10.1186/s12885-016-2761-8. PMID 27629548